CLINICAL TRIAL: NCT04457947
Title: Exploring an Aromatherapy Intervention in an Acute Care Setting
Brief Title: Exploring Aromatherapy Intervention in Acute Care
Acronym: Aromatherapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Amanda Bulette Coakley, principal investigator, Massachusetts General Hospital
Other Study IDs: 2019-P002663
Record Dates: First submitted 2020-03-06; First posted 2020-07-07 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Pregnant Women; Surgical Patients
Keywords: aromatherapy; lavendar; ginger

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to explore how the use of inhaled essential oils impacts the experience of a laboring and postoperative surgical patient. It is expected that the aromatherapy intervention will decrease levels of nausea, anxiety, and improve the perception of being cared for in laboring mothers and patients recovering from surgery. By learning more about aromatherapy, the investigators may be able to expand the aromatherapy intervention to more patients in other Massachusetts General Hospital departments.

20 laboring patients will be recruited on admission to the labor and delivery inpatient unit. They will be invited to participate in this study by nurses caring for them.

20 postoperative surgical patients will be recruited on admission to the surgical inpatient unit. They will be invited to participate in this study by nurses caring for them

DETAILED DESCRIPTION:
Aromatherapy is a complementary integrative intervention that can be incorporated into nursing care to optimize health. It is defined as the use of essential oils, obtained from aromatic plants, for therapeutic properties. Most State Boards of Nursing recognize clinical aromatherapy as part of holistic nursing. There are benefits of using aromatherapy for nausea, comfort, wellbeing, perception of care and anxiety which are common symptoms associated with hospitalized patients.

Hospitalized patients often report a myriad of symptoms and increasingly ask for alternative ways to manage them. According to the National Center for Complementary and Integrative Health (NCCIH), a national survey in the United States. Four national surveys report that a third or more of US adults routinely use complementary and alternative medicine (CAM) therapies (e.g. chiropractic, massage, yoga, supplements, acupuncture) to treat their principal medical conditions with total expenditures exceeding $34 billion in 2007. A global shift in healthcare is moving toward wider acceptance of a philosophical value-guided health approach that includes a whole-person/whole-system caring healing health perspective . Complementary therapies have become more widely known and used in western healthcare. The human consciousness shift toward wellness is allowing models and possibilities of inner healing and emotional and mental health.

Despite widespread use and acceptance of complementary therapies in community settings, there is some resistance to implementing such strategies in the acute care setting. There are no reports of randomized clinical trials supporting such interventions in acute care settings. Some evidence exists to support some complementary and integrative interventions.

One intervention that is cost effective and non-invasive is aromatherapy. While research indicates that the use of aromatherapy has been effective in managing nausea, anxiety, and discomfort, there are limited rigorous studies supporting its use in the acute care setting. More work is needed to understand if aromatherapy is a feasible intervention to implement in the acute care setting. Further research is needed to explore which essential oils are most effective for symptom management in patients in the acute care setting.

Two groups of patients that commonly report anxiety, discomfort and nausea are postoperative surgical patients and laboring obstetric patients. This study will explore the use of aromatherapy as an intervention used by nurses to assist laboring obstetric patients and postoperative elective surgical patients manage symptoms of nausea, anxiety, and discomfort. Aromatherapy will serve as an adjunct and not as a replacement for standard routine care.

For many women, having a baby provides their first experience as a patient in a hospital setting. Many women are hesitant to utilize pharmacological methods to decrease pain, anxiety, and nausea associated with their labor experience due to fear of harming their baby. As such, women increasingly turn to complementary therapies such as aromatherapy as a means of retaining control over their childbirth experience. Odor has a direct pathway to the limbic part of the brain, in particular to the amygdala that governs fear. Familiar smells such as lavender may be calming and soothing at stressful times such as during childbirth. Surgery is another stressful time for patients.

Much of the limited research on aromatherapy is two decades old. A British evaluative study of 8,058 mothers delivering in a large teaching hospital between 1990 and 1998 indicated that lavender aromatherapy relieved feelings of anxiety and fear (61%), pain (6%), improved contractions (6%), reduced feelings of nausea and vomiting (14%) and improved general well-being (7%). Lavender, frankincense and rose were found to relieve anxiety in labor. There is some evidence that aromatherapy has been successfully used by midwives to reduce the level of anxiety during the antepartum period. In a clinical randomized trial of 100 women in labor, the level of anxiety of women in both the intervention (P=0.03) and control (P=0.003) groups after the intervention was reduced after the intervention. Findings from these studies also indicate that there were minimal to no side effects.

Post-operative nausea and vomiting (PONV) continue to be a major cause of patient dissatisfaction affecting hospitalized patients. Although conventional approaches can be very effective in managing PONV, some patients are intolerant of drug side effects or decline use the medications. There is some evidence that inhalation of lavender, ginger, peppermint and other oils are alternative techniques that have been used successfully with postoperative patients in helping to manage discomfort and nausea. It is suggested that aromatherapy can be tried before conventional techniques in managing nausea and vomiting and used alongside it in a complementary manner.

This quasi experimental mixed method study will utilize a convenience sample and a pre- and post-study design study to determine the feasibility of implementing an aromatherapy intervention on two acute care units.

Primary outcomes for this study include anxiety, nausea, perception of caring and well-being. In addition, an open-ended qualitative inquiry will be used to further explore the experience including potential positive and negative outcomes.

This study will be conducted on two acute care inpatient care areas: labor delivery unit with healthy pregnant women and on a general adult surgical unit with persons having elective surgery. Twenty patients will be recruited from the surgical unit and thirty from the obstetrical unit.

Study Procedure Using inclusion/exclusion outlined criteria below, all patients meeting inclusion criteria will be introduced to the aromatherapy intervention by the nurse research assistant who is caring for them. Potential participants will be asked if they wish to enroll in the study during their hospitalization. If they express interest, patients will be given information regarding the investigation and the informed consent form to read. The Principal Investigator (PI) will be notified. The nurse research assistant will answer any questions of the potential participant and if the patient agrees to enroll in the study, the nurse research assistant will obtain a written informed consent. Once enrolled, demographic variables will be collected and the following measures will be obtained before the aromatherapy intervention and immediately after the intervention.

1. Vital signs including blood pressure, pulse and level of respirations
2. Generalized Anxiety Disorder (GAD-7) scale
3. Visual Analog Scale (VAS) for nausea
4. Watson Caritas Patient Score
5. Warwick-Edinburgh mental well-being scale (WEMWBS)

The day after the inhaled essential oil is administered, a different member of the study team will ask the patient open-ended questions about their experience with aromatherapy.

Aromatherapy intervention

* Lavender inhaled essential oil will be used for perceived caring, wellbeing and reported anxiety in all patients
* Ginger essential oil will be used for patients who report nausea.
* A certified study clinician will administer the inhaled essential oil during labor or during the postoperative recovery period.

Patients on the labor and delivery inpatient unit (Blake 14) and post-operative surgical inpatient unit (Ellison 7) will be offered aromatherapy as an alternative treatment for nausea and anxiety in labor and during the post-operative surgical recovery period.

Aromatherapy is an integrative, nonpharmacological intervention that will be explored as a treatment of nausea, vomiting, anxiety, and comfort in labor and post-operative surgical recovery.

On admission, the patient will be asked to list their allergies. If the patient has allergies to study aromatherapy oils, then the patient will be excluded from the study. If the patient appears to develop an allergic reaction or any other adverse reaction to an administered essential oil, the use of aromatherapy in this patient will be discontinued immediately and the patient will be removed from the study.

All patients on Labor & Delivery and on Ellison 7 will be asked if they wish to participate in this investigation. Patients must be at least 18 years of age and able to provide informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatient Blake 14 and Ellison 7
2. Able to give consent

Exclusion Criteria:

1. Patients who have allergies or sensitivities to essential oils, lavender and ginger 2. Patients with bleeding or clotting disorder 3. Patients who are unable to give informed consent 4. Patients who are younger than 18 years old 5. Patients who are unable to read or write English

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 mothers in labor 20 patients who have undergone surgical operation
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
1. To understand the impact of aromatherapy on wellbeing as measured by the Warwick-Edinburgh mental well-being scale . | through study completion, an average six months
  Measures well-being, 14 items with a 5 point likert scale, 1=none of the time and 5=all of the time
2. To understand the impact of aromatherapy on perception of caring as measured by the Watson Caritas Patient Score | through study completion, an average six months
  Assess patient perspective on compassionate care with a 7 point likert scale, 1= never, 7= always

OTHER OUTCOMES:
3. To understand the impact of aromatherapy on anxiety as measured by Generalized Anxiety Disorder (GAD-7) scale | through study completion, an average six months
  Measuring anxiety. A score of 10 or higher means significant anxiety is present
4. To understand the impact of aromatherapy on nausea as measured by VAS for nausea. | through study completion, an average six months
  Measuring nausea. s a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measure.s a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measure. is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. It is a meaurement instrument for subjective characteristics. ! being low and 10 being high
1. To qualitatively explore the overall experience of patients who have had an aromatherapy intervention | through study completion, an average six months
  Understanding the experience of aromatherapy through qualitative open ended questions

CONTACTS AND LOCATIONS:
Overall Officials: Amanda B Coakley, PhD, Principal Investigator — Massachusetts General Hospital

REFERENCES:
- [Result] Brewer BB, Watson J. Evaluation of Authentic Human Caring Professional Practices. J Nurs Adm. 2015 Dec;45(12):622-7. doi: 10.1097/NNA.0000000000000275. PMID 26502069
- [Result] Rashidi-Fakari F, Tabatabaeichehr M, Mortazavi H. The effect of aromatherapy by essential oil of orange on anxiety during labor: A randomized clinical trial. Iran J Nurs Midwifery Res. 2015 Nov-Dec;20(6):661-4. doi: 10.4103/1735-9066.170001. PMID 26793249
- [Result] Buckle J. Literature review: should nursing take aromatherapy more seriously? Br J Nurs. 2007 Jan 25-Feb 7;16(2):116-20. doi: 10.12968/bjon.2007.16.2.22772. PMID 17353823
- [Result] Burns EE, Blamey C, Ersser SJ, Barnetson L, Lloyd AJ. An investigation into the use of aromatherapy in intrapartum midwifery practice. J Altern Complement Med. 2000 Apr;6(2):141-7. doi: 10.1089/acm.2000.6.141. PMID 10784271
- [Result] Eisenberg DM, Kaptchuk TJ, Post DE, Hrbek AL, O'Connor BB, Osypiuk K, Wayne PM, Buring JE, Levy DB. Establishing an Integrative Medicine Program Within an Academic Health Center: Essential Considerations. Acad Med. 2016 Sep;91(9):1223-30. doi: 10.1097/ACM.0000000000001173. PMID 27028029